CLINICAL TRIAL: NCT00919230
Title: Randomised Trial Comparing Iron Supplementation Versus Placebo in the Treatment of Anaemia After Hip Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Collaborators: Peterborough Hospitals Hip Fracture Project (Unknown)
Responsible Party: Principal Investigator, Martyn J Parker, research fellow, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R&D/2003/21
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Hip Fracture
Keywords: Hip fracture; iron therapy; anaemia
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no treatment (No Intervention): no iron given
- ferrous sulphate (Experimental): iron given
  Interventions: Drug: Ferrous sulphate tablets

INTERVENTIONS:
Drug: Ferrous sulphate tablets — 200mg twice daily for four weeks
  Arms: ferrous sulphate

SUMMARY:
At present our current practice is to provide a course of oral iron therapy for those patients with a post-operative haemoglobin which is below normal, but not severe enough to require a blood transfusion. Such a practice is not without side effects from the iron tablets, namely ingestion, nausea, diarrhoea, constipation. There is little evidence in the literature to support the current practice of using iron, with only one small randomised trial suggesting such therapy is unnecessary. We propose to recruit 300 patients recovering from a hip fracture with a post-operative haemoglobin below 11g/l. For those patients willing to enter the study, half will be given oral iron therapy (ferrous sulphate 200mg twice daily) for one month. The haemoglobin will be checked when the patients attends the hip fracture clinic at 6 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients with anaemia after surgery for a hip fracture

Exclusion Criteria:

* absence of anaemia, inability to provide consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
6 week hemoglobin | 6 weeks after surgery

SECONDARY OUTCOMES:
Length of hospital stay side effects of therapy mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Parker, Principal Investigator — Peterborough Hospitals
Locations (1):
- Peterborough city hospital, Peterborough, Cambs, United Kingdom

REFERENCES:
- [Background] Parker MJ. Iron supplementation for anemia after hip fracture surgery: a randomized trial of 300 patients. J Bone Joint Surg Am. 2010 Feb;92(2):265-9. doi: 10.2106/JBJS.I.00883. PMID 20124051